CLINICAL TRIAL: NCT02990624
Title: Effect of Photochemotherapy on Cardiometabolic Markers in Patients With Psoriasis With and Without Atherosclerosis
Brief Title: Cardiovascular Risk Evaluation in Psoriasis Treated With Photochemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Vanessa Suzanne Galal Hafez, Lecturer of dermatology, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVR in UV phototherapy
Record Dates: First submitted 2016-11-29; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Psoriasis Vulgaris
Keywords: psoriasis; photochemotherapy; atherosclerosis; metabolic syndrome; cardiovascular risk
MeSH Terms: conditions — Psoriasis; Atherosclerosis; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High risk group (Active Comparator): Patients with psoriasis and atherosclerosis will receive PUVA therapy for 36 sessions divided as 3 sessions weekly
  Interventions: Radiation: PUVA
- Low risk group (Active Comparator): Patients with psoriasis but no atherosclerosis detected, will receive PUVA therapy for 36 sessions divided as 3 sessions weekly
  Interventions: Radiation: PUVA
- Control group (No Intervention): Age-matching apparently normal individuals will receive no interventions but will perform investigational tests.

INTERVENTIONS:
Radiation: PUVA — 36 sessions of psoralen-ultraviolet A, divided as 3 sessions weekly
  Arms: High risk group; Low risk group

SUMMARY:
Ultraviolet (UV) phototherapy is a standard treatment for many inflammatory dermatological diseases, including psoriasis. The systemic effects of UV phototherapy are still not well studied. There are several factors that may affect patient's cardiovascular (CV) risk during UV phototherapy. Atherosclerosis is now known to have an inflammatory origin and to be frequently associated with psoriasis. In this study the investigators aim at studying the effect of psoralen-UVA phototherapy on several biomarkers of CV risk in patients with psoriasis with or without atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Disease affecting > 10% body surface area
* Patient willing to commit to 3 sessions weekly for 3-6 months without interruption

Exclusion Criteria:

* Disease severity less than 10% body surface area
* Patients unable to commit for therapeutic schedule due to work or residence issues.
* pregnant and lactating females
* photosensitive dermatoses

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Comparative change in photoinduced oxidation and related change in cardiovascular risk between both risk groups in response to photochemotherapy | day 0 to end of 12 weeks (end of 36 sessions, 3 sessions weekly of photochemotherapy) and/or clinical cure whichever comes first
  Comparison between both risk groups in the amount of change between baseline level and end of study level of oxidized low density lipoprotein

SECONDARY OUTCOMES:
comparative number of patients with metabolic syndrome after therapy in both groups | end of 12 weeks (end of 36 sessions, 3 sessions weekly of photochemotherapy) and/or clinical cure whichever comes first
  Comparison between both risk groups as regards the number of patients with metabolic syndrome
Comparative changes in metabolic syndrome component 1: waist circumference | day 0 to end of 12 weeks (end of 36 sessions, 3 sessions weekly of photochemotherapy) and/or clinical cure whichever comes first
  Comparison between both risk groups in the amount of change between baseline level and EOS level of waist circumference
Comparative changes in metabolic syndrome component 2: arterial blood pressure | day 0 to end of 12 weeks (end of 36 sessions, 3 sessions weekly of photochemotherapy) and/or clinical cure whichever comes first
  Comparison between both risk groups in the amount of change between baseline level and EOS level of arterial blood pressure
Comparative changes in metabolic syndrome component 3: blood sugar | day 0 to end of 12 weeks (end of 36 sessions, 3 sessions weekly of photochemotherapy) and/or clinical cure whichever comes first
  Comparison between both risk groups in the amount of change between baseline level and EOS level of blood sugar
Comparative changes in metabolic syndrome component 4: serum lipids | day 0 to end of 12 weeks (end of 36 sessions, 3 sessions weekly of photochemotherapy) and/or clinical cure whichever comes first
  Comparison between both risk groups in the amount of change between baseline level and EOS level of serum lipids
Atherosclerotic changes in the high risk group in response to PUVA | end of 12 weeks (end of 36 sessions, 3 sessions weekly of photochemotherapy)
  comparison of duplex arteriography findings in the high risk group between before and after treatment
Correlation between cutaneous response and systemic response to photochemotherapy in both risk groups | day 0 to end of 12 weeks (end of 36 sessions, 3 sessions weekly of photochemotherapy) and/or clinical cure whichever comes first
  Correlation between PASI score after treatment and other parameters of systemic response (hs-CRP, ox-LDL, metabolic syndrome components)

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology department - faculty of medicine- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No